CLINICAL TRIAL: NCT04609384
Title: The Effect on a Timer-device on the Time Spend on Surgical Rub
Brief Title: Nudging Effect of Timer on Surgical Rub
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sygehus Lillebaelt (Other)
Responsible Party: Principal Investigator, per hviid gundtoft, Principal Investigator, MD, PhD, Sygehus Lillebaelt
Other Study IDs: PHG_1_timer
Record Dates: First submitted 2020-06-30; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Operation Wound; Infection; Bacterial Infections; Surgical Procedure, Unspecified
MeSH Terms: conditions — Surgical Wound Infection; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prior to installation of device: Health care workers who perform the surgical rub prior to installation of the device that should increase the time spend on surgical rub.
  Interventions: Device: Alcohol rub timer device
- Post device installation: Health care workers who perform the surgical rub following installation of the device that should increase the time spend on surgical rub.
  Interventions: Device: Alcohol rub timer device

INTERVENTIONS:
Device: Alcohol rub timer device — A device that should help the surgeon to increase the time spend on surgical rub. Further detail cannot be described due to confidence

SUMMARY:
To study whether a device has a nudging effect on the time spend on surgical rub.

DETAILED DESCRIPTION:
The investigators observed the time spend on surgical rub prior to an operation. The investigators do not record names, age, sex or orther features about the health care workers who perform the surgical rub.

After 200 observations a device will be attach to the dispenser that might help increase the time spend on the surgical rub in the operathing theather. The investigatos will then make another 200 observations to see if the device cause an increase in the time spend on surgical rub.

ELIGIBILITY:
Inclusion Criteria:

• All professional health care workers, who perform surgical ru

Exclusion Criteria:

* Students and other persons at a hospital, who are not paid to be working at the hospital.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All health care workers who perform alcohol rub.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Time | Seconds used on surgical rub at least 300 seconds. Observation begin from start of surgical rub (defined as the time when the dispenser is activated) to the end of surgical rub (defined as the time when the surgeon pick up the surgical gown)
  time used on surgical rub

CONTACTS AND LOCATIONS:
Locations (1):
- Sygehus Lillebaelt, Kolding, Denmark

IPD SHARING:
Plan to Share IPD: No
We do not keep indivicual participants data but treat all data anonymous.